CLINICAL TRIAL: NCT03522311
Title: Evaluation of 25-gauge Vitrectomy Surgical Outcomes for Proliferative Diabetic Retinopathy by Preoperative Glycemic Control and Renal Function
Brief Title: Surgical Outcomes for Proliferative Diabetic Retinopathy by Preoperative Glycemic Control and Renal Function
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Department of Ophthalmology, Kyorin University
Other Study IDs: Kyorineye025
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
The surgical outcomes of 25-gauge vitrectomy for proliferative diabetic retinopathy has been evaluated by preoperative glycemic control and renal function

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the surgical outcomes of 25-gauge vitrectomy for proliferative diabetic retinopathy by preoperative glycemic control and renal function.

ELIGIBILITY:
Inclusion Criteria:

* The patients had25-gauge vitrectomy for proliferative diabetic retinopathy

Exclusion Criteria:

* The patients had hemodialysis , followed up less than 6 months, had vitrectomy for diabetic macular edema and macular ration but not macular detachment.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eyes with proliferative diabetic retinopathy
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Visual acuity measurement | 6 months
  Visual acuity improvement from baseline

SECONDARY OUTCOMES:
Presence of postoperative vitreous hemorrhage | 6 months
  Incidence of postoperative vitreous hemorrhage

OTHER OUTCOMES:
Presence of postoperative retinal detachment | 6 months
  Incidence of postoperative retinal detachment

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center

IPD SHARING:
Plan to Share IPD: No